CLINICAL TRIAL: NCT06557291
Title: Relapse-Free Survival With Adjuvant Dabrafenib/Trametinib Therapy After Relapse on Adjuvant Checkpoint Inhibitor Therapy and Subsequent Surgical Resection in Patients With BRAF V600-mutated Stage III/IV Melanoma
Brief Title: Relapse-Free Survival With Adjuvant Dabrafenib/Trametinib Therapy in Patients With BRAF V600-mutated Stage III/IV Melanoma
Status: Completed | Type: Observational
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: CTMT212AUS65
Record Dates: First submitted 2024-08-13; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: BRAF V600 Mutated-Stage III/IV Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Dabrafenib and Trametinib Combination Therapy Cohort: Adult BRAF V600 patients with resected stage III/IV melanoma that relapsed during or after CPI as their first adjuvant therapy and were again rendered free of disease and received adjuvant dab/tram combination therapy.

SUMMARY:
This was a retrospective chart review study of all proto-oncogene B-Raf (BRAF) V600-mutated patients who received adjuvant checkpoint inhibitor (CPI) therapy, relapsed locoregionally or distantly, and were again resected to no evidence of disease (NED) and treated with adjuvant dabrafenib and trametinib (dab/tram) combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Any patient at least 18 years of age at the time of diagnosis of stage III/IV melanoma.
* Received surgical resection with no residual disease following initial stage III/IV melanoma diagnosis.
* Documented local or central assay-positive for tumor BRAF V600E/K mutation.
* Received adjuvant CPI alone or in combination with any other immune treatment as their first adjuvant therapy.
* Following adjuvant CPI, relapsed (locoregionally or distantly) on or off treatment and was again rendered free of disease after subsequent surgical resection.
* Received additional adjuvant dab/tram combination therapy after failing adjuvant CPI and being subsequently resected to NED.

Exclusion Criteria:

* Previous administration of any BRAF- or mitogen-activated protein kinase (MEK)-targeted therapies.
* More than 120 days duration between surgery to render the patient NED after relapsing during or after adjuvant CPI therapy and initiation of dab/tram adjuvant therapy.
* Administration of any intervening antitumor medical and/or radiation therapy between failing adjuvant CPI and initiation of adjuvant dab/tram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2023-11-16 (Actual)

PRIMARY OUTCOMES:
Relapse-free Survival-2 (RFS-2) | Up to 63 months
  RFS-2 was defined as the time from the study index date until the date of the earliest clinician-documented disease progression, death, or start of a new line of anticancer treatment due to disease progression. Patients without a progression event as described above were censored at the last available follow-up, defined as last known clinic visit or last known contact with the patient (if occurred outside the clinic setting).
  Index date was defined as the date that dab/tram combination therapy was initiated after being rendered disease-free for a second time following additional resection after prior relapse on initial CPI adjuvant therapy.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 63 months
  OS was defined as the time from the study index date until death due to any cause. Patients without a death event were censored at last available follow-up, defined as last known clinic visit or last known contact with the patient (if occurred outside the clinic setting).
  Index date was defined as the date that dab/tram combination therapy was initiated after being rendered disease-free for a second time following additional resection after prior relapse on initial CPI adjuvant therapy.
Distant Metastases-free Survival (DMFS) | Up to 63 months
  DMFS was defined as the time from the study index date until the first observation of disease progression with distant metastasis. Patients without a DMFS event as described above were censored at last available follow-up, defined as last known clinic visit or last known contact with the patient (if occurred outside the clinic setting).
  Index date was defined as the date that dab/tram combination therapy was initiated after being rendered disease-free for a second time following additional resection after prior relapse on initial CPI adjuvant therapy.
Number of Patients with an Adverse Event (AE) Related to Dabrafenib and Trametinib Combination Therapy | Up to 63 months
Mean Number of Times an AE Related to Dabrafenib and Trametinib Combination Therapy was Experienced | Up to 63 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States